CLINICAL TRIAL: NCT03821376
Title: Correlation of Contrast Enhanced Ultrasound of Renal Masses With Pathologic Grade: A Prospective Comparison of Quantitative and Qualitative Findings
Brief Title: Correlation of Renal Mass Pathologic Grade and Contrast Enhanced Ultrasound (CEUS)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped due to staffing issues that impacted ability to recruit.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jordan K. Swensson, Assistant Professor of Clinical Radiology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1901057253
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Renal Malignant Tumor
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Imaging findings for enrolled patients will be compared to pathologic grading
Masking Description: Imaging reviewers will be blinded to pathologic grade
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Renal malignancy (Experimental): Patients with renal mass(es) identified by cross sectional imaging, specifically ultrasound following the intravenous injection of Lumason
  Interventions: Drug: Contrast enhanced ultrasound with Lumason

INTERVENTIONS:
Drug: Contrast enhanced ultrasound with Lumason — Following consent, they will undergo contrast enhanced ultrasound of their known renal mass(es). This will be performed at University hospital following intravenous administration of Lumason (2.5 mL per injection, maximum of 2 injections per mass).
  Other Names: Ultrasound

SUMMARY:
Patients with renal lesions suspicious for renal cell carcinoma (RCC) have a variety of different treatment pathways available to them. Imaging surveillance is being used frequently on smaller renal masses, and radiologists are being asked to biopsy more renal lesions to better guide decision making by urology. This is in large part due to the pathologic grade of renal masses having been shown to correlate with patient outcomes. The World Health Organization (WHO) or Fuhrman grade is the standard grading scale used by pathologists for RCC. The goal of this study will be to correlate contrast enhanced ultrasound findings with the pathologic grade of RCC. Specifically, the investigators hypothesize that tumors with different pathologic grades will show different patterns of qualitative enhancement, as well as different perfusion kinetics.

DETAILED DESCRIPTION:
Renal malignancies are relatively common, with lifetime risk ranging from 1 in 48 in men to 1 in 83 in women, of which RCC is the most common. RCC comes in a variety of subtypes, and pathologic grade has been shown to be one factor that correlates with patient prognosis [Novara et al]. The most commonly used pathologic grading systems are the WHO or Fuhrman scale, which rely on histologic features of the tumor such as nuclear size, irregularity, and nucleolar prominence.

Care of patients with RCC depends on a number of factors, including size and pathologic grade. As such, radiologic surveillance with CT and MRI is common, and percutaneous biopsy of renal masses for the purpose of pathologic grading is also relatively common. While percutaneous biopsy of renal masses is the least invasive way to obtain tissue, these still carry risks, especially of hemorrhage give the vascular nature of the kidneys and RCC.

Contrast enhanced ultrasound has been shown to have the ability to differentiate renal masses from normal background renal parenchyma [Barr et al]. It has the unique ability to be used in patients with renal dysfunction as it is excreted by the liver and lungs. As such, it is well suited for use in patients with underlying renal pathology. This study will aim to use contrast enhanced ultrasound to evaluate the qualitative and quantitative features of renal masses prior to surgical removal, and then evaluate for correlation of these features with pathologic grading following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Previously identified renal mass with radiology and clinical features consistent with RCC
* Clinical care plan includes partial or total nephrectomy

Exclusion Criteria:

* Less than 18 years of age
* Currently pregnant
* Renal mass with clinical care plan that does not include nephrectomy
* Renal mass suspected to be non RCC neoplasm by imaging and clinical data
* Renal mass unable to be visualized by grayscale ultrasound
* Known renal vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Swennson, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Renal Malignancy
Started | 12
Completed | 9
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Renal Malignancy
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Lesion pathology [Number; unit: participants] — Renal pathologic grading done following WHO grading system for renal cell carcinoma (RCC). Lesions may be considered grade 1-4, with 4 representing the most aggressive pathology appearance. Kidney lesions that are not RCC are not given a grade.
  participants
    WHO grade 2 lesion | 6
    WHO grade 3 lesion | 1
    Oncocytoma | 2

OUTCOME MEASURES:

1. Primary Outcome: Contrast Enhanced Ultrasound Features of Renal Masses (Time to Peak, Mean Transit Time)
Description: Ultrasound images will be reviewed for quantitative post contrast features (time to peak, mean transit time)
Time Frame: 6 months
Population: 9 patients who completed enrollment and proceeded to surgery; staffing and software issues precluded acquisition of quantifiable ultrasound data on all but 1 of the patients who proceeded to surgery
Measure: Number; unit: seconds
Arm/Group | Renal Malignancy
Number analyzed (Participants) | 1
seconds
  Time to peak enhancement (seconds) | 4.76
  Mean transit time (seconds) | 32.1

2. Primary Outcome: Contrast Enhanced Ultrasound Features of Renal Masses (Peak Intensity)
Description: Ultrasound images will be reviewed for quantitative post contrast features. Specifically peak intensity, which is measured in "enhancement units." A higher value represents more blood flow to the renal mass.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: enhancement units
Arm/Group | Renal Malignancy
Number analyzed (Participants) | 1
enhancement units | 2.26

ADVERSE EVENTS:
Time Frame: From enrollment to time of surgery (2 months)
Arm/Group | Renal Malignancy
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03821376/Prot_SAP_001.pdf